CLINICAL TRIAL: NCT07251361
Title: SENSORFIT-4HEART: Smart Exercise preScriptiOn and Remote Monitoring FITness Platform for HEART Failure With Preserved Ejection Fraction
Brief Title: Effects of a Multicomponent Training Program on Cardiac Function, Skeletal Muscle Metabolism, Functional Capacity, and Quality of Life in Patients With HFpEF: SENSORFIT-4HEART Study
Acronym: SENSORFIT-4HEA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: NavarraBiomed Biomedical Research Center (Other); Centro de Investigación Médica Aplicada (CIMA) (Unknown); Complejo Hospitalario de Navarra (Other); Instituto de Investigación Sanitaria de Navarra (IdiSNA) (Unknown)
Responsible Party: Principal Investigator, Dr Mikel Izquierdo, Principal Investigator, Universidad Pública de Navarra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PI_2023/146; PI_2023/146 (Other: Fundación Miguel Servet)
Record Dates: First submitted 2025-09-23; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Exercise; PeakVO2; Cardiac function; Skeletal muscle bioenergetics; Quality of life; Exerkines
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise program (Experimental): Participants assigned to this arm will receive supervised multicomponent exercise program delivered twice per week, combining resistance training (RT) with aerobic training within the same session. The RT session duration will increase progressively from 10 to 20 min at 40-70 % of one repetition maximum (1-RM) twice weekly. RT include progressively three series × 10-15 repetitions of leg press, knee extensors, chest press, and horizontal rowing.
  Interventions: Behavioral: Supervised training
- Usual care (No Intervention): Patients allocated to this arm will receive the usual care plus explicit recommendations for home-based aerobic and strength training (Vivifrail program).

INTERVENTIONS:
Behavioral: Supervised training — Supervised training
  Arms: Supervised exercise program

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a complex syndrome with increasing incidence and poor prognosis, accounting for up to 50% of heart failure cases. It is strongly associated with aging, cardiovascular risk factors (hypertension, diabetes, obesity), and is more prevalent in women than men. Patients with HFpEF frequently present with dyspnea, debilitating fatigue, poor quality of life, frequent hospitalizations, and high mortality rates. This study aims to evaluate the effects of a structured exercise program on cardiac function, skeletal muscle metabolism, functional capacity, and quality of life in patients with HFpEF, and to explore whether these benefits are mediated by circulating exerkines.

DETAILED DESCRIPTION:
Standard pharmacological treatments have shown limited prognostic benefit, highlighting the need for non-pharmacological strategies. Exercise training may represent an effective therapeutic tool, with potential to improve cardiac remodeling, skeletal muscle bioenergetics, exercise tolerance, and quality of life. Importantly, exerkines-molecules secreted by skeletal muscle and other organs in response to exercise-may mediate systemic beneficial effects by modulating metabolic, immuno-inflammatory, and growth pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure with preserved ejection fraction according to 2021 ESC guidelines for Heart Failure.
* Left ventricular ejection fraction (LVEF) >40%, and/or evidence of structural and/or functional cardiac abnormality (diastolic dysfunction, elevated filling pressures, BMI>30 kg/m2)
* Elevated natriuretic peptides (BNP ≥35 pg/mL or NT-proBNP ≥125 pg/mL)
* Stable symptomatic heart failure patients (New York Heart Association functional class II-III/IV) during the last month

Exclusion Criteria:

* Participation in cardiac rehabilitation within the past 12 months.
* Contraindications to physical exercise training.
* Alternative diagnoses that could explain symptoms of HF (dyspnea, fatigue), in the judgment of the cardiologist.
* Significant pulmonary disease, including primary pulmonary hypertension.
* Severe chronic lung disease, including COPD requiring home oxygen, chronic nebulizer therapy, long-term oral steroids, or hospitalization for decompensated pulmonary disease within the past 12 months.
* Hemoglobin <10 g/dL.
* Body mass index (BMI) >40 kg/m².
* Inability to perform a valid baseline cardiopulmonary exercise test
* Inability to comprehend study information or complete questionnaires (e.g., psychiatric disorder, dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption | Baseline and 12-week
  Changes in peak oxygen consumption between and within groups at 12-week Unit of measure of peak oxygen consumption: mL/kg/min. Maximal functional capacity will be evaluated using incremental and symptom-limited cardiopulmonary exercise testing on a bicycle ergometer, beginning with a workload of 25 W and increasing gradually in a ramp protocol at 25-W increments every 3 minute. We define maximal functional capacity as when the patient stops pedalling because of symptoms and the respiratory exchange ratio (RER) was >1. Gas exchange data and cardiopulmonary variables were averages of values taken every 10 seconds. Peak oxygen consumption (PeakVO2) was defined as the highest value of VO2 during the last 20 seconds of exercise.

SECONDARY OUTCOMES:
Lean mass (kg) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Changes in blood pressure | Baseline and 12-week
  Systolic and diastolic blood pressure of participants in fasting condition will be analyzed by electronic tensiometer and reported in mmHg.
Changes in Heart rate | Baseline and 12-week
  Heart rate of participants in fasting condition will be analyzed by electronic tensiometer and reported in pulses/min.
Changes in muscle strength | Baseline and 12-week
  Grip strength of participants will be measured using a manual dynamometer and reported in kg. Pectoral press, bilateral leg-press, knee extension, and back press) will be measured using a eGYM machines and reported in kg
Changes in quality of life | Baseline and 12-week
  We will use the EuroQol five-dimension five-level questionnaire (EQ-5D-5L) to assess health-related quality of life. The EQ-5D-5L includes five domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each rated on a 5-point scale ranging from 1 (no problems) to 5 (extreme problems). The responses are combined into an index value ranging from -0.594 to 1, where higher scores indicate a better health-related quality of life.
Physical activity and sedentary behaviour (in minutes) | Baseline and 12-week
  Physical activity level objectively measured using Actigraph Accelerometry. This will be worn on the waist and will passively record physical activity and sedentary behavior.
Pittsburgh Sleep Quality Index | Baseline and 12-week
  A 19-item self-report questionnaire that assesses subjective sleep quality and disturbances over the past month will be evaluated by Pittsburgh Sleep Quality Index. The global score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Epidemiological Studies-Depression Scale questionnaire | Baseline and 12-week
  Depression levels will be assessed using the Center for Epidemiological Studies-Depression Scale (CES-D) questionnaire, which is validated and widely employed in cardiometabolic patients. The CES-D consists of 20 items, each rated on a 4-point Likert scale ranging from 0 (rarely or none of the time) to 3 (most or all of the time), assessing the frequency of depressive symptoms during the past week. The total score ranges from 0 to 60, with higher scores indicating greater depressive symptomatology.
Cognitive Function | Baseline and 12-week
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a validated screening tool that evaluates multiple cognitive domains, including executive function, memory, attention, language, and visuospatial abilities. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance.
Adherence to the Mediterranean Diet | Baseline and 12-week
  Adherence to the Mediterranean dietary pattern will be assessed using the Mediterranean Diet Adherence Screener (MEDAS), a validated 14-item questionnaire designed to evaluate compliance with key components of the Mediterranean diet. Each item is scored 0 or 1, depending on whether the dietary criterion is met, yielding a total score ranging from 0 to 14, where higher scores indicate greater adherence to the Mediterranean diet.
Psychological Distress | Baseline and 12-week
  The Kessler Psychological Distress Scale (K10) will be used to assess nonspecific psychological distress, including symptoms of anxiety and depression, experienced over the past four weeks. The K10 consists of 10 items, each rated on a 5-point Likert scale ranging from 1 (none of the time) to 5 (all of the time), resulting in a total score between 10 and 50. Higher scores indicate greater psychological distress.
Haematology | Baseline and 12-week
  Erythrocyte count (×10⁶ cells/µL), haematocrit (%), haemoglobin (g/dL), platelet count (×10³ cells/µL), leukocyte count (×10³ cells/µL), and erythrocyte mean corpuscular volume (fL) will be quantified using a Coulter haematology analyzer (Brand, City, Country).
Concentrations of circulating cytokines, adipokines, myokines, and bone metabolism biomarkers. | Baseline and 12-week
  Plasma concentrations of pro-inflammatory and anti-inflammatory cytokines (IL-1β, IL-2, IL-6, IL-8, IL-10, IFN-γ, TNF-α, IL-1ra, and TNF sRII-α), adipokines (adiponectin, adipsin, resistin, PAI-1 active, insulin, and leptin), and myokines (irisin) will be quantified using Luminex xMAP technology. In addition, biomarkers related to bone metabolism (ACTH, DKK-1, FGF-23, osteocalcin, osteopontin [OPN], osteoprotegerin, PTH, and sclerostin [SOST]) will be measured with the same platform. Each analyte will be reported separately as an independent outcome, with concentrations expressed in pg/mL or ng/mL, as appropriate for the specific biomarker.
Resting energy expenditure | Baseline and 12-week
  Resting energy expenditure is measured in the fasting and fed state by indirect calorimetry
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | Baseline and 12-week
  N-terminal pro-B-type natriuretic peptide (NT-proBNP) will be quantified by standardized immunoassay (e.g., electrochemiluminescence immunoassay, ECLIA) following manufacturer's instructions
Lean mass index (kg/m2) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Appendicular lean mass index (kg/m2) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass index (kg/m2) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass (kg) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Visceral adipose tissue (kg) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Lean mass/fat mass ratio | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat free mass | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Whole bone mineral density (g/cm2) | Baseline and 12-week
  Dual-energy X-ray absorptiometry (DXA) body composition measure

OTHER OUTCOMES:
Lipidomic | Baseline and 12-week
  Lipidomic will be expressed and analyzed in plasma and serum according to their intensity measured in arbitrary units (UA), which carries a direct relation with its concentration in blood. Performed in a randomly selected sub-sample of approximately 30% of study participants
Mitochondrial leak respiration | Baseline and 12-week
  Mitochondrial O2 flux is measured by high-resolution respirometry in muscle mass tissue. Performed in a randomly selected sub-sample of approximately 30% of study participants
Proteome profile | Baseline and 12-week
  Assessment of changes in proteins profile following intervention in blood. Performed in a randomly selected sub-sample of approximately 30% of study participants. Each outcome will be reported separately, with concentrations expressed in pg/mL or ng/mL, as appropriate for the specific analyte.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pública de Navarra (UPNA), Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No